CLINICAL TRIAL: NCT01159691
Title: A Multicentric, Non-interventional Study on Switching From Oral Parkinson Therapy to Neupro® in Patients With Idiopathic Parkinson's Disease With Gastrointestinal Symptoms
Brief Title: Change in Gastrointestinal Complaints After Switch From Oral Parkinson's Disease Treatment to Neupro® Transdermal Patch
Acronym: NON-GI
Status: Completed | Type: Observational
Sponsor: UCB Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: SP0970
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro®; Parkinson's disease; Gastrointestinal; Switch from oral therapy to patch
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neupro: Routine treatment as per approved label in Europe/ in accordance with the terms of the local marketing authorization for Neupro® transdermal patch.

SUMMARY:
The study intends to collect data on gastrointestinal symptoms (swallowing disorders, heartburn, feeling of fullness, nausea, vomiting, abdominal pain, diarrhea) and on patient satisfaction under everyday practice conditions after changing treatment to Neupro® transdermal patch in patients suffering from idiopathic Parkinson´s Disease with gastrointestinal symptoms while being treated with oral antiparkinson drugs. The objective of the study is to ascertain whether switching therapy to Neupro® transdermal patch can provide any relief in gastrointestinal symptoms.

DETAILED DESCRIPTION:
Routine treatment as per approved label in Europe in accordance with the terms of the local marketing authorization for Neupro®.

ELIGIBILITY:
Inclusion Criteria:

* The decision to prescribe Neupro® must have been made by the physician before and independently of his/her decision to include the patient in the study
* The patient's treatment must be in accordance with the terms of the local marketing authorization (MA) for Neupro®
* The patient must have a diagnosis of Idiopathic Parkinson's disease
* The patient must have signed the Consent form regarding study information, data transfer and use
* Patient suffering from gastrointestinal symptoms while being treated with oral Parkinson's medication

Exclusion Criteria:

Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's Disease (PD) suffering from gastrointestinal complaints under oral anti-parkinson treatment; treated in Germany by neurological outpatient centers (clinic/ practice of neurologist).
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (21):
- Germany (21):
  - 02, Berlin
  - 24, Bochum
  - 38, Buchholz
  - 7, Cologne
  - 30, Erbach im Odenwald
  - 14, Gera
  - 28, Göttingen
  - 16, Karlstadt am Main
  - 40, Lauf an der Pegnitz
  - 39, Lüneburg
  - 37, München
  - 31, Neuburg am Inn
  - 35, Nuremberg
  - 22, Schriesheim
  - 34, Schwäbisch Gmünd
  - 21, Stadtroda
  - 12, Stuttgart
  - 36, Stuttgart
  - 1, Ulm
  - 32, Ulm
  - 29, Wolfratshausen

REFERENCES:
- [Derived] Woitalla D, Kassubek J, Timmermann L, Lauterbach T, Berkels R, Grieger F, Muller T. Reduction of gastrointestinal symptoms in Parkinson's disease after a switch from oral therapy to rotigotine transdermal patch: a non-interventional prospective multicenter trial. Parkinsonism Relat Disord. 2015 Mar;21(3):199-204. doi: 10.1016/j.parkreldis.2014.11.024. Epub 2014 Dec 4. PMID 25595315
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in June 2010 in order to end up with 21 centers in Germany.
Pre-assignment Details: 76 patients were included in the Enrolled Set (ES), 75 of whom were treated with Neupro® at least once during the Observational Period and, thus, constituted the Safety Set (SS). The Full Analysis Set (FAS) encompassed all 65 patients who had been treated with Neupro® at least once and who had valid Baseline and Follow-up Visit values.
Period: Overall Study
Arm/Group | Neupro
Started | 76
Completed | 54 (Multiple discontinuation reasons were possible.)
Not Completed | 22
Not completed — Lost to Follow-up | 2
Not completed — Unknown reasons | 1
Not completed — Discontinued Neupro due to Adverse Event | 6
Not completed — Discontinued Neupro due to other reasons | 1
Not completed — Disc. Neupro other & lost to follow-up | 2
Not completed — Disc. Neupro other & unknown reasons | 7
Not completed — Disc. Neupro due to AE & unknown reasons | 2
Not completed — Disc. Neupro lack of efficacy & unknown | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics show the Enrolled Set (ES). ES encompasses those patients who have been included in this study and for whom data are available on the first Visit (initial examination).
Arm/Group | Neupro
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 70.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 45
Region of Enrollment [Number; unit: participants]
  Germany | 76
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 78.1 (12.9)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.1 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 3 in the Assessment of Intensity of Gastrointestinal (GI) Complaints for Any Reason as Per Visual Analogue Scale (VAS)
Description: Patients were asked to classify the intensity of their GI complaints on a scale ranging from 0 (no complaints) to 100 (extremely severe complaints). Negative values indicate an improvement from Baseline to Visit 3 with larger negative values showing a better improvement.
Time Frame: From Baseline to Visit 3 (approximately 6 weeks)
Population: Of the 65 subjects in the Full Analysis Set, 58 are included in this analysis.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Neupro
Number analyzed (Participants) | 58
millimeter (mm) | -26.8 (28.8)

2. Primary Outcome: Change From Baseline to Visit 3 in the Sum Score of Gastrointestinal (GI) Complaints
Description: Sum score of GI complaints was calculated from frequency and intensity of the complaints. The intensity of GI complaints during the last week ranges from 0 (no complaints) to 3 (severe) and the frequency of these complaints during the last week ranges from 0 (never) to 4 (every day).
  For each of the seven GI complaints assessed at a visit (swallowing disorders, heartburn, feeling of fullness, nausea, vomiting, abdominal pain, and diarrhea), intensity and frequency were multiplied to achieve individual item scores of GI complaints (range: 0 - 12).
  Finally, the sum score of GI complaints per visit was calculated by accumulating 6 of the 7 item scores (excluding swallowing disorders, which was recorded at Baseline only) for patients with valid values in each score (range: 0 - 72). Negative values indicate an improvement from Baseline to Visit 3 with larger negative values showing a better improvement.
Time Frame: From Baseline to Visit 3 (approximately 6 weeks)
Population: Of the 65 subjects in the Full Analysis Set, 58 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro
Number analyzed (Participants) | 58
units on a scale | -8.4 (8.1)

3. Primary Outcome: Assessment of Patient Satisfaction Referring to Gastrointestinal (GI) Complaints Following Treatment Switch to Neupro® at Visit 2
Description: Patient satisfaction referring to GI complaints is classified into 5 categories:
  * Missing
  * Very satisfied
  * Satisfied
  * Moderately satisfied
  * Not satisfied.
Time Frame: At Visit 2 (after approximately 2-4 weeks)
Population: All of the 65 subjects in the Full Analysis Set are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Neupro
Number analyzed (Participants) | 65
participants
  Missing | 1
  Very satisfied | 25
  Satisfied | 26
  Moderately satisfied | 8
  Not satisfied | 5

4. Primary Outcome: Assessment of Patient Satisfaction Referring to Gastrointestinal (GI) Complaints Following Treatment Switch to Neupro® at Visit 3
Description: as for outcome 3
Time Frame: At Visit 3 (after approximately 6 weeks)
Population: All of the 65 subjects in the Full Analysis Set are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Neupro
Number analyzed (Participants) | 65
participants
  Missing | 7
  Very satisfied | 28
  Satisfied | 22
  Moderately satisfied | 6
  Not satisfied | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the entire Study Period from Baseline (Visit 1) up to approximately 6 weeks (Visit 3).
Description: Adverse Events refer to the Safety Set. The Safety Set encompasses all included patients who were treated with Neupro® at least once. Of the 76 patients in the Enrolled Set, 75 patients are included in the Safety Set.
Arm/Group | Neupro
Serious Adverse Events (participants affected / at risk) | 4/75
Other Adverse Events (participants affected / at risk) | 21/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro (N=75)
Death (General disorders) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Haematoma evacuation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro (N=75)
Lacrimation increased (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Application site erythema (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Drug ineffective (General disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
On and off phenomenon (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days